CLINICAL TRIAL: NCT03650673
Title: A Prospective Cohort Study of Patients Suffering From Hand Osteoarthritis
Brief Title: A Prospective Cohort Study of Patients Suffering From Hand Osteoarthritis Symptoms
Acronym: COARDIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RECHMPL17_0391; 2017-A03378-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-08-22; First posted 2018-08-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hand Osteoarthritis
Keywords: Hand osteoarthritis; Prospective cohort; Cartilage; Mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Test: Identification of subgroups of patients with (Other)
  Interventions: Diagnostic Test: Identification of subgroups of patients with early AD with risk of progression

INTERVENTIONS:
Diagnostic Test: Identification of subgroups of patients with early AD with risk of progression — Clinical examination with questionnaires, Biological collection, Imaging (radiography, densitometry, ultrasound, and MRI)

SUMMARY:
The late-stage forms of degenerative osteoarthritis (OA) are very debilitating and less affordable to therapy. The main objective is to identify early onset symptoms of hand OA patients through imaging techniques (such as ultrasound and MRI). Our primary endpoint is to specify patients with high risk of radiological profression (X-ray).

ELIGIBILITY:
Inclusion Criteria:

- Early digital osteoarthritis must combine the clinical AND radiological definition.

Clinical definition:

At least one of the following 4 criteria: Pain or stiffness or swelling or deformity of a digital joint (IPP and / or IPD) A breach of at least one PPI and / or IPD Age under 60 at the time of the first symptoms Clinical symptoms have been changing for less than 3 years

Radiographic definition:

The presence of the achievement of at least one PPI and / or IPD. Presence of at least two of the following three criteria: pinching, marginal subchondral condensation, marginal osteophyte Erosion on radiography is not an exclusion criteria

- Consent form signed

Exclusion criteria:

* patients suffering from rheumatoid arthritis, rheumatoid psoriasis or any other inflammatory rheumatism
* patients suffering from metabolic diseasis such as gout, hemochromatosis, Wilson's disease; or from congenital disease such as displasie, osteogenesis,
* Presence of advanced radiographic osteoarthritis based in Kellgreen Lawrence score (=4) in one joint among the 10 previous sites.
* Not able to provide a sample of blood for any reasons
* MRI contraindication
* Being in exclusion period determined by another previous study
* Subject non affiliated to social insurance
* Pregnant or lactating women
* Vulnerable people based in L1121-5 article of CSP
* Elderly subject or protected subjects disabled to give their consent
* Subjects private of freedom by court or administrative order

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression judged by the number of joints whose KL index has evolved | 2 years
  Evaluation of prognostic role of imaging factors in x-ray progression of early onset hand osteoarthritis

SECONDARY OUTCOMES:
The number of painful / swollen or deformed joints in the hands. | 2 years
  Photographs of the patients' hands will be taken at each visit.
The location of painful / swollen or deformed joints in the hands. | 2 years
  Photographs of the patients' hands will be taken at each visit.
The intensity of pain over the last 48 hours | 2 years
  The intensity of pain over the last 48 hours will be assessed by the patient at each visit on a visual analogue scale (VAS). EVA pain (visual analogue scale over 100 mm): one-dimensional measurement of the intensity of pain. EVA pain is a continuous scale consisting of a horizontal line from 0 (no pain) to 100 mm (maximum pain)
The activity of the disease over the last 48 hours | 2 years
  The activity of the disease over the last 48 hours will be evaluated at each visit by the patient and the doctor on a visual analog scale from 0 (no pain) to 100 mm (maximum pain)
The aesthetic impact of osteoarthritis of the hands | 2 years
  The aesthetic impact of osteoarthritis of the hands will be evaluated at each visit by the patient on a visual analog scale from 0 (no pain) to 100 mm (maximum pain)
The number of consumption of care in the month preceding the visit | 2 years
The number of hand surgery during follow-up 56/5000 The number of a hand surgery during follow-up | 2 years
The grip force measured by a dynamometer | 2 years
The impact on pain and function on the hand measured by the AUSCAN questionnaire | 2 years
  The impact on pain and function measured by the AUSCAN questionnaire. This is a functional index including 15 questions with a specific orientation to osteoarthritis of the hands, assessing pain / stiffness and function. The score varies from 0 to 60. Fill in the questionnaire: 7 min
The impact on pain and function on the hand measured by the COCHIN functional index | 2 years
  The impact on pain and function measured by the COCHIN functional index wich is oriented towards AD. It includes 18 questions, ranging from 0 to 5, and is particularly interested in the impact of osteoarthritis of the hands on the daily activities (cooking, clothing, hygiene, office ...) of the patient. The score varies from 0 to 90. Questionnaire filling time: 5 min
The impact on pain and function on the hand measured by a 6-minute walk test | 2 years
  The impact on pain and function measured by a 6-minute walk test that characterizes an overall assessment of functional ability to exercise. The patient is asked to walk as much as possible for 6 minutes (round trip in a 30m corridor), the pace of walking is freely chosen (ATS Recommendations, 2002)
The impact on pain and function measured the IPAQ International Physical Activity Questionnaire | 2 years
  The short version with 7 questions will be used
The professional impact measured by the WPAI questionnaire which measures the deficiencies of paid work and unpaid work over the last 7 days | 2 years
  The WPAI questionnaire is an instrument for measuring deficiencies in paid work and unpaid work over the last 7 days. It measures absenteeism, presenteeism as well as the deficiencies of unpaid activity due to a health problem. It contains 6 questions and has already been used during AD
Impact on quality of life measured by the Health Assessment Questionnaire (HAQ) | 2 years
  The Health Assessment Questionnaire (HAQ) is a measure of quality of life in health. The questionnaire is designed to be completed by the patient himself, without the help of a doctor. We will use an adaptation of the HAQ, the Modified Health Assessment Questionnaire (MHAQ), as in the Kwok et al. Study, with 8 questions about the function of the hand. The score ranges from 0 to 3. The average score reported in osteoarthritis studies is 0.8. It is 0.49 in the global population.
The impact on the quality of life measured by the SF-36 questionnaire | 2 years
  The SF-36 questionnaire assesses the quality of life. It is a validated international questionnaire. It consists of 36 items evaluating 8 dimensions. It can be used in health economics studies as a variable in the calculation of a Quality Adjusted Life Year (QALY) to determine the cost-effectiveness of a health intervention. Fill in the questionnaire: 10 min.
The impact on the quality of life measured by the EQ-5D-3L questionnaire (https://euroqol.org) | 2 years
  This score varies between 0 and 1: 0 represents death, and 1 the best quality of life possible. So, this score indicates the decrease in quality of life compared to an optimal state of health. The more desirable a health state, the higher the score associated with it. Negative scores are possible if the subject perceives a state of health worse than death. The EQ-5D-3L includes the following five dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Each dimension has 3 levels: absence of problems, presence of problems and extreme problems. Questionnaire filling time: 5 min
The Impact on Quality of Life Measured by the Michigan Hand Outcome Questionnaire (MHQ) | 2 years
  It is an international questionnaire validated with 6 items, which assesses the aesthetic impact of osteoarthritis of the hands. The questionnaire includes the function of the overall hand, the activities of daily life, the pain, the work, the appearance of the hands and the satisfaction of the patient with the functionality of his hands. In the ladder pain, a high score indicates more intense pain, while in the rest of the items, a better score reveals better hand functionality. Duplicate filling time: 15 min.
The psychological impact of pain measured by the HAD questionnaire (Hospital Anxiety and Depression) | 2 years
  This questionnaire assesses the psychological impact of the patient. It consists of 14 questions with 4 possible answers. This score makes it possible to differentiate a level of anxiety and a level of depression according to the answers. Each sub-scale varies from 0 to 21. Questionnaire filling time: 5 min
The aesthetic impact of osteoarthritis of the hands with the Michigan Hand Outcome Questionnaire | 2 years
  The aesthetic impact of osteoarthritis of the hands will be evaluated at each visit by the patient with the help of the Michigan Hand Outcome Questionnaire. It is an international questionnaire validated with 6 items, which assesses the aesthetic impact of osteoarthritis of the hands. The questionnaire includes the function of the overall hand, the activities of daily life, the pain, the work, the appearance of the hands and the satisfaction of the patient with the functionality of his hands. In the ladder pain, a high score indicates more intense pain, while in the rest of the items, a better score reveals better hand functionality. Duplicate filling time: 15 min (MHQ)

CONTACTS AND LOCATIONS:
Overall Officials: Yves-Marie PERS, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of Rheumatology, CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No